CLINICAL TRIAL: NCT00735228
Title: Benefit of Tight Glycemic Control in Surgical Patients: Prospective Randomized Clinical Trial
Brief Title: Tight Glycemic Control by Artificial Pancreas
Acronym: KMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kochi University (Other)
Collaborators: Oita University (Other); University of Tokushima (Other)
Responsible Party: Kochi Medical School, Kochi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCAP0802; Kochi Medical School
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Last update posted 2008-08-18 (Estimated); Status verified 2008-08

CONDITIONS: Pancreatic Disease; Cardiovascular Diseases
Keywords: surgery; artificial pancreas; tight glycemic control; Liver
MeSH Terms: conditions — Pancreatic Diseases; Cardiovascular Diseases | interventions — Pancreas, Artificial; Insulin Infusion Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Perioperative blood glucose was controlled within the normal levels (80-110 mg/dL) by artificial pancreas.
  Interventions: Device: Artificial pancreas
- 2 (Active Comparator): Perioperative blood glucose concentration was controlled within the range from 140 to 160 mg/dL by artificial pancreas.
  Interventions: Device: Artificial pancreas

INTERVENTIONS:
Device: Artificial pancreas — Artificial endocrine pancreas (NIKKISO Company)
  Other Names: artificial endocrine pancreas (NIKKISO Company)

SUMMARY:
Hyperglycaemia has been repeatedly associated with risk of mortality and morbidity in the intensive care unit (ICU). The evidence currently available is in favour of a 'normal ≤ 6.1 mmol/l' level for blood glucose control in ICUs according to two large randomized control trials of Van den Berghe G and is not supportive of J. Miles's viewpoint in this debate. In this study, the investigators would like to evaluate that the target of blood glucose level, whether is a normal level (80-110 mg/dL) or another level (140-160 mg/dL), should be set for the reduction of perioperative mortality and complications.

DETAILED DESCRIPTION:
Our previous prospective randomized clinical trial suggested that the postoperative morbidities were reduced by tight glycemic control of a normal level for blood glucose using artificial pancreas. However, the most feared one is hypoglycaemia, which, when severe and prolonged, may cause convulsions, coma and brain damage, as well as cardiac arrhythmias. Recently, Ven den Berghe G report that the development of accurate, continuous blood glucose monitoring devices, and preferably closed-loop systems for computer-assisted blood glucose control in the ICU, will help to avoid hypoglycaemia. In our study, no hypoglycemia showed in more than 100 patients who performed perioperative tight glycemic control by artificial pancreas.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were suffering from liver, pancreas or cardio-vascular diseases, were informed of the purpose and details of the study, and written consent was obtained from them prior to enrolment.

Exclusion Criteria:

* Patient exclusion criteria included a body weight loss greater than 10% during the six months prior to surgery
* The presence of distant metastases, or seriously impaired function of vital organs due to respiratory, renal or heart disease.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2008-08; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
The incidence of hypoglycemia | during hospitalization

SECONDARY OUTCOMES:
The incidence of postoperative infectious complications and calculate the total costs during hospitalization | during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Takehiro Okabayashi, MD, PhD, Study Director — Kochi Medical School
Locations (1):
- Kochi Medical School, Nankoku, Japan

REFERENCES:
- [Derived] Okabayashi T, Shima Y, Sumiyoshi T, Kozuki A, Tokumaru T, Iiyama T, Sugimoto T, Kobayashi M, Yokoyama M, Hanazaki K. Intensive versus intermediate glucose control in surgical intensive care unit patients. Diabetes Care. 2014 Jun;37(6):1516-24. doi: 10.2337/dc13-1771. Epub 2014 Mar 12. PMID 24623024